CLINICAL TRIAL: NCT04072107
Title: Epstein-Barr Virus DNA to Systemic Therapy for Treatment Adaptation in High Risk Nasopharyngeal Carcinoma (EP-STAR Trial) A Phase II, Multi-center, Biomarker-guided, Umbrella Trial
Brief Title: EPstein-barr Virus DNA Response to Systemic Therapy for Treatment Adaptation in High Risk NPC (EP-STAR)
Acronym: EP-STAR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: National Cancer Centre, Singapore (Other); Wuzhou Red Cross Hospital (Other); First People's Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Ying Sun, Vice president, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2019-185-01
Record Dates: First submitted 2019-08-24; First posted 2019-08-28 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma; EBV DNA; Biomarker-guided; Treatment adaptation
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — sintilimab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Experimental): Patients receive GP IC + IMRT concurrent with cisplatin chemotherapy + capecitabine AC. All patients will receive concurrent cisplatin (100 mg/m2) every 3 weeks, in a total of three cycles. All patients will receive low-dose metronomic capecitabine (650 mg/m2 bid, oral, d1-21, q3w) until disease progression, or intolerable toxicity or 6 months.
  Interventions: Drug: Capecitabine
- Arm II (Experimental): Patients receive GP IC + IMRT concurrent with cisplatin chemotherapy and anti-PD-1 therapy (sintilimab) + anti-PD-1 therapy (sintilimab) AC. All patients will receive concurrent cisplatin (100 mg/m2) and sintilimab (200 mg, IV drop 30-60 min) every 3 weeks in a total of three cycles. All patients will receive adjuvant anti-PD-1 therapy (sintilimab, 200 mg, IV drop 30-60 min, q3w) in a total of nine cycles until disease progression, or intolerable toxicity or 6 months.
  Interventions: Drug: sintilimab

INTERVENTIONS:
Drug: sintilimab — Investigate whether capecitabine would be able to improve prognosis in patients at high risk groups
  Arms: Arm II
Drug: Capecitabine — Investigate whether capecitabine would be able to improve prognosis in patients at intermediate risk groups
  Arms: Arm I

SUMMARY:
The investigators aim to investigate whether incorporating on-treatment EBV DNA surveillance for monitoring tumor responses to treatment and for guiding individuliased treatment adaptation can improve prognosis in nasopharyngeal carcinoma patient . For patients with detectable EBV DNA after one cycle of IC, which then drops to undetectable levels during the following IC cycles (intermediate responders/intermediate relapse risk), the investigators aim to investigate whether additional adjuvant metronomic capecitabine would benefit this subgroup. For patients with detectable EBV DNA after three cycles of IC or with EBV DNA bounce during the induction phase (insensitive to IC/high relapse risk), the investigators aim to investigate whether concurrent administration of anti-PD-1 therapy during the following treatment phases (including concurrent phase and adjuvant phase) can benefit this subgroup.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is a unique head and neck cancer characterized by an extremely unbalanced global distribution. The highest incidence is observed in endemic regions, such as southern China and Southeast Asia, with an age-standardized rate of 3.0 per 100,000 in China to 0.4 per 100,000 in Caucasian populations. The fast progress of modern imaging and the application of intensity-modulated radiotherapy (IMRT) has improved the local control rate significantly. Distant metastasis has become the major cause of treatment failure.

The 2018 National Comprehensive Cancer Network (NCCN) guideline recommends concurrent chemoradiotherapy (CCRT) ± induction chemotherapy (IC)/adjuvant chemotherapy (AC) as the standard treatment for stage II-IVa disease (category 2A). While it is worth noting that there is extensive heterogeneity among patients with NPC, and even among patients with the same disease stage, the risk of relapse varies. More importantly, patients can have differing sensitivity to RT and chemotherapy. The abovementioned reasons result in over-treatment in some patients with relatively low relapse risk; intensive treatments lead to unnecessary toxicities, and greatly affect quality of life (QoL). On the other hand, the current treatment strategy may be not optimal for patients with high relapse risk or who are not sensitive to traditional chemoradiotherapy. Therefore, there is an urgent need for identifying and applying promising biomarkers, real-time monitoring of patient responses to treatment, predicting relapse risk, and guiding real-time treatment adaptation for individualized therapy.

The investigators aim to investigate whether incorporating on-treatment EBV DNA surveillance for monitoring tumor responses to treatment and for guiding individuliased treatment adaptation can improve prognosis in nasopharyngeal carcinoma patient . For patients with detectable EBV DNA after one cycle of IC, which then drops to undetectable levels during the following IC cycles (intermediate responders/intermediate relapse risk), the investigators aim to investigate whether additional adjuvant metronomic capecitabine would benefit this subgroup. For patients with detectable EBV DNA after three cycles of IC or with EBV DNA bounce during the induction phase (insensitive to IC/high relapse risk), the investigators aim to investigate whether concurrent administration of anti-PD-1 therapy during the following treatment phases (including concurrent phase and adjuvant phase) can benefit this subgroup.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed, pathologically proven World Health Organization (WHO) type II/III untreated LANPC;
2. LANPC (except T3N0, according to the 8th edition of the AJCC/UICC clinical staging system);
3. Age at diagnosis: 18-65 years;
4. Eastern Cooperative Oncology Group (ECOG) score: 0-1
5. Receiving recommended three cycles of induction chemotherapy (IC) (gemcitabine-cisplatin [GP] regimen);
6. Pre-treatment and post-IC1 cell-free Epstein-Barr virus (cfEBV) DNA > 0 copy/mL; systemic cfEBV DNA monitoring during IC phase for risk stratification;
7. Normal hematic, liver, and kidney function: hemoglobin (HG) > 90 g/L; neutrophil > 1.5 × 109/L; platelet > 100 × 109/L; total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 2.5 × ULN; alkaline phosphatase (ALP) ≤ 2.5 × ULN; creatinine clearance (Ccr) ≥ 60 mL/min;
8. Female subjects capable of becoming pregnant agree to use reliable contraceptive measures from screening to 1 year after treatment;
9. Patients will be required to sign informed consent forms and be willing and able to comply with the requirements for visits, treatment, laboratory tests, and other research requirements stipulated in the research schedule.

Exclusion Criteria:

1. Receiving surgery, target therapy, and/or immunotherapy during or before induction phase;
2. Hepatitis B surface antigen-positive [HBsAg(+)],hepatitis B virus (HBV) DNA > 1×103 copy/mL; hepatitis C virus (HCV) antibody(+);
3. Other previous or concurrent malignant tumors, except adequately treated non-melanoma skin cancer, cervical carcinoma in situ, and thyroid papillary cancer;
4. Pregnant or lactating women (a pregnancy test should be considered for fertile women with an active sex life);
5. Previously treated with radical radiotherapy (RT), except non-melanoma skin cancers outside intended RT treatment volume;
6. Uncontrolled heart disease, e.g.: 1) Heart failure, Hew York Heart Association (NYHA) level ≥ 2; 2) unstable angina; 3) myocardial infarction in the past 1 year; 4) supraventricular or ventricular arrhythmia requiring treatment or intervention;

   *For patients recruited to Arm II, the additional exclusion criteria are:
7. Active, known, or suspected autoimmune disease (including, but not limited to, uveitis, enteritis, hepatitis, pituitary, nephritis, vasculitis, hyperthyroidism, hypothyroidism, and asthma requiring bronchiectasis). Exceptions are type I diabetes mellitus, hypothyroidism requiring hormone replacement therapy, and skin disorders requiring no systemic treatment (e.g., vitiligo, psoriasis, alopecia);
8. Received live vaccine within 1 month before treatment initiation;
9. Allergy to macromolecular protein preparations, or any component of sintilimab;
10. Human immunodeficiency virus (HIV)-positive or diagnosed with Acquired Immune Deficiency Syndrome (AIDS).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival | 2 year
  FFS will be measured from the day of enrollment until treatment failure, death from any cause, or the last follow-up visit, whichever occurred first.

SECONDARY OUTCOMES:
overall survival | 2 year
  measured from the day of enrollment until death due to any cause, or the last follow-up visit.
Distant metastasis failure-free survival | 2 year
  measured from the day of enrollment until death until distant metastasis , or the last follow-up visit.
Locoregional failure-free survival | 2 year
  measured from the day of enrollment until death until local and/or regional recurrence, or the last follow-up visit.
Adverse events | up to 5 years
  The incidence of immune-related and other adverse events
Patient reported quality-of-life score | up to 2 years
  Patient reported quality of life would be evaluated using the Quality of Life Questionnaire-Core 30 module (QLQ-C30)
Biomarker analysis | Through study completion
  Exploratory biomarker analysis that would be able to predict patient treatment benefits, for example PD-L1 expression, tumor mutational burden, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Sun, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Currently, there is no plan to make individual participant data (IPD) available to other researchers.